CLINICAL TRIAL: NCT05846334
Title: A MHealth Intervention to Reduce Perceived Stress in Patients with Ischemic Heart Disease
Brief Title: MHealth Intervention to Reduce Perceived Stress in Patients with Ischemic Heart Disease
Acronym: mStress-IHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Collaborators: Universität Duisburg-Essen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-11015-BO
Record Dates: First submitted 2023-03-27; First posted 2023-05-06 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-05

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Device: mindfulHeart
- Control group (No Intervention)

INTERVENTIONS:
Device: mindfulHeart — 'mindfulHeart' is an interactive, self-guided and patient-oriented mHealth intervention for the reduction of stress in patients with IHD and includes automated feedback via visualization of changes in patient reported outcome measures (PROMs).
  Arms: Intervention group

SUMMARY:
Stress is highly prevalent in patients with ischemic heart disease (IHD) and is associated with lower health-related quality of life and worsened cardiovascular outcome. The importance of stress management is now recognized in recent cardiovascular guidelines. However, effective stress management intervention are not implemented in clinical routine yet. The development of easily disseminated eHealth interventions, particularly mHealth, may offer a cost-effective and scalable solution to this problem. The aim of the proposed trial is to assess the efficiency and cost-effectiveness of the mHealth intervention 'mindfulHeart' in terms of reducing stress in patients with IHD.

DETAILED DESCRIPTION:
Chronic stress occurs over an extended period, from months to years, and can result in several adverse health consequences. The relationship between chronic stress and cardiovascular diseases continues to be subject of extensive research. Recent large studies have shown that chronic stress is linked to heightened risk for cardiovascular diseases (CVD), leading to its recognition in current clinical guidelines. Chronic stress was demonstrated as risk factor for the development, but also for the progression of CVD, and research has found associations between stress measurements and traditional cardiovascular risk factors. Stress is also considered as relevant player in the pathophysiological cascade of coronary atherosclerosis formation (e.g., inflammatory response, endothelial dysfunction, platelet aggregation) until the development of clinical apparent ischemic heart disease (IHD). Measures of stress have been associated with the onset and progression of further cardiovascular disorders, like coronary calcification, atrial fibrillation, and stroke. In patients with IHD, stress has also been implicated as an acute trigger of myocardial ischemia and infarction, malignant arrhythmias, and sudden cardiac death.

Although the body of evidence examining the stress-IHD connection is growing, there continues to be a lack of recognition of this association in clinical practice and of effective and scalable interventions. Desirable would be the sustainable integration of targeted therapy in cardiology practice that involves screening for stress, referral to psychological, and/or behavioral therapy or to other stress reducing interventions (e.g. meditation, holistic self-care programs, or other complementary approaches). Although ongoing group support and concomitant coaching in other lifestyle-related fields such as diet and exercise are conductive to long-term adherence, the establishment of area-wide structured stress management programs is resource-intensive and currently not available.

A potential solution to cost-prohibitive stress reduction programs is the development of easily disseminated eHealth intervention, which can be effective and scalable, and easier to implement in the context of a busy clinical practice. The term "eHealth" encompasses a wide range of electronic solutions, such as mobile phones (mHealth) and computers that can enhance and broaden the scope of medical care.

Especially mHealth interventions are perceived to offer several advantages that may overcome some of the limitations of face-to-face approaches, including anonymity, 24/7 availability, reduced costs in terms of traveling to courses for both participants and instructors, high scalability, and a low access threshold. Enabling participants to be reached earlier than in classical face-to-face trainings, such interventions may have the potential to prevent even the onset of more severe chronic stress or mental health problems. The effectiveness of eHealth interventions for stress reduction was shown in a recent meta-analysis.

The link between stress and increased mortality and morbidity in CVD is obvious and includes also an undeniable reduction in health-related quality of life (HRQoL). This lead to the fact that the search for novel therapeutic strategies is inevitable. Therefore, the investigators aim in the current study to evaluate the efficacy and cost-effectiveness of the digital stress management intervention 'mindfulHeart' in terms of sustainable stress reduction in the target population.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of IHD
* elevated perceived stress for at least 4 weeks
* own an Internet-enabled smartphone and know how to use it
* have provided written informed consent

Exclusion Criteria:

* Participants who have severe cognitive impairment and/or communication difficulties that may affect their ability to participate in the study
* psychiatric or medical conditions that require alternative treatment
* no private internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
combined global stress measure | 3 months, after intervention
  The outcome is based on a published RCT in Circulation by Blumenthal et al. [34]. A global stress measure (mean rank), was the primary outcome combining the following components at baseline and following treatment: Beck Depression Inventory II, Spielberger Anxiety Inventory-State, General Health Questionnaire, PROMIS Anger Questionnaire, and Perceived Stress Scale. A range from 1 to 147 was present with higher scores suggestive of better function. The change in each individual scaled score is presented in primary outcome 2. (see also NCT00981253)

SECONDARY OUTCOMES:
Health-related quality of life | Baseline, after 3 months, after 4 months, after 6 months, after 9 months, after 15 months
  we will apply two instrument to measure health-related quality of life. Namely the Short Form-36 health questionnaire and the European Quality of Life 5 Dimensions 5 Level survey (EQ-5D-5L) [36,37]. The SF-36 is an eight-dimensional scale consisting of 36 items. It assesses health-related quality of life based on physical, social, and psychological functioning, role behavior due to physical and psychological functional impairment, physical pain, general health perception, and vitality. The EQ-5D-5L consists of five health-related dimensions that can be assessed at five levels. In addition, the questionnaire contains a visual analog scale for assessing general health
Disease-specific effect of angina on patients' physical function and quality of life | Baseline, after 3 months, after 4 months, after 6 months, after 9 months, after 15 months
  We will also include the Seattle Angina Questionnaire (SAQ). The 7-item version of the SAQ is a shortened version of the original 19-item SAQ and has been shown to be highly valid, reliable, and sensitive to clinical change. These ranges of SAQ scores are strongly and independently correlated with the risk of subsequent death, the risk of myocardial infarction, and health care costs
Changes in functional capacity | Baseline, after 3 months, after 4 months, after 6 months, after 9 months, after 15 months
  changes in functional capacity will be recorded using the established 6-minute walk test
Blood pressure | Baseline, after 3 months, after 4 months, after 6 months, after 9 months, after 15 months
  To evaluate the effect of the intervention on blood pressure , this parameters will be assessed with the average of three consecutive measurements at rest. The standard measurement approach was always performed in the same quiet room at a consistent controlled temperature and after a resting period of at least 20 minutes. The same examination sequence was maintained for all study subjects. To obtain reliable measurements, the patients were asked not to speak and to lie quietly during the entire measurement.
Heart rate | Baseline, after 3 months, after 4 months, after 6 months, after 9 months, after 15 months
  To evaluate the effect of the intervention on heart rate , this parameters will be assessed with the average of three consecutive measurements at rest. The standard measurement approach was always performed in the same quiet room at a consistent controlled temperature and after a resting period of at least 20 minutes. The same examination sequence was maintained for all study subjects. To obtain reliable measurements, the patients were asked not to speak and to lie quietly during the entire measurement.
Self-efficacy | Baseline, after 3 months, after 4 months, after 6 months, after 9 months, after 15 months
  To evaluate self-efficacy, we will utilize the Generalized Self-Efficacy Scale (GSES) in its German version [41]. The GSES is a self-administered questionnaire that measures an individual's optimistic self-beliefs and self-efficacy in dealing with challenging demands and stressful events in life. Each of the 10 items is rated on a 4-point Likert scale.
combined global stress measure | Baseline, after 3 months, after 4 months, after 6 months, after 9 months, after 15 months
  The outcome is based on a published RCT in Circulation by Blumenthal et al. [34]. A global stress measure (mean rank), was the primary outcome combining the following components at baseline and following treatment: Beck Depression Inventory II, Spielberger Anxiety Inventory-State, General Health Questionnaire, PROMIS Anger Questionnaire, and Perceived Stress Scale. A range from 1 to 147 was present with higher scores suggestive of better function. The change in each individual scaled score is presented in primary outcome 2. (see also NCT00981253)
Depression symptoms (BDI-II) | Baseline, after 3 months, after 4 months, after 6 months, after 9 months, after 15 months
  The BDI-II is a self-report questionnaire comprising 21 items that assess depression severity. Its reliability and validity have been established through various studies among diverse populations and cultural backgrounds. Higher scores indicates increased depression symptoms
Anxiety symptoms (STAI) | Baseline, after 3 months, after 4 months, after 6 months, after 9 months, after 15 months
  The STAI is the most authoritative tool for assessing anxiety in adults, precisely distinguishing between transient "state anxiety" and persistent "trait anxiety". The STAI measures anxiety with 20 items and has a range of 20 to 80. A higher score indicates more pronounced anxiety
PROMIS-Anger Scale | Baseline, after 3 months, after 4 months, after 6 months, after 9 months, after 15 months
  The PROMIS Anger scale comprises eight items that evaluate various aspects of anger. Scores on the scale range from 8 to 40, with higher scores indicating greater levels of anger
GHQ | Baseline, after 3 months, after 4 months, after 6 months, after 9 months, after 15 months
  The GHQ assesses general distress and consists of 12 items. Respondents' scores range from 0 to 36, where higher scores correspond to increased distress
Perceived Stress Scale | Baseline, after 3 months, after 4 months, after 6 months, after 9 months, after 15 months
  The Perceived Stress Scale-10 item version is a short tool for the assessment of how individuals perceive stress in their lives. The values range from 0 to 40. Higher values indicate higher perceived stress [46].
  (l) In-treatment assessments: at the start of each intervention module (weekly), the following assessment instruments will be applied: Distress Thermometer (DT), Patient Health Questionnaire-4 (PHQ-4) and self-generated measures to assess coping skills and self-efficacy

OTHER OUTCOMES:
Treatment satisfaction | Baseline, after 3 months, after 4 months, after 6 months, after 9 months, after 15 months
  the adapted German version of the Client Satisfaction Questionnaire for Internet-based interventions (CSQ-I) is an 8-item assessment instrument that evaluates participants' overall satisfaction with the intervention. Responses are measured on a 4-point Likert scale.
Usability | Baseline, after 3 months, after 4 months, after 6 months, after 9 months, after 15 months
  The System Usability Scale is used to assess the usability of the intervention, which is a 10-item questionnaire rated on a 5-point Likert scale. To determine the perceived usefulness of our healthcare smartphone app, we will also use a healthcare smartphone app evaluation survey. Responses are measured on a 4-point Likert scale.
Predictors of usage behavior | Baseline, after 3 months, after 4 months, after 6 months, after 9 months, after 15 months
  assessing the predictors of actual usage behavior is crucial as interventions can only benefit patients who use them. Therefore, it is important to evaluate the predictors of uptake for the intervention. In order to do so, the Unified Theory of Acceptance and Use of Technology and it modified questionnaire will be applied [52].
Cost-effectiveness | after 15 months
  the objective of conducting an economic evaluation is to assess the cost-effectiveness of the intervention from the viewpoint of payers. This evaluation will involve a cost-effectiveness analysis and will be calculated based on the EQ-5D-5L questionnaire.
Cost-utility | after 15 months
  To determine the cost-utility, quality-adjusted life years will be calculated based on the EQ-5D-5L questionnaire. The resource utilization will be evaluated by means of a questionnaire and will be measured in monetary units using the established standards of health economics. Furthermore, the costs per reduced unit of stress are assessed and compared between the intervention group and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Lortz, MD, Principal Investigator — University of Duisburg-Essen
Locations (1):
- Westdeutsches Herz- und Gefäßzentrum, Klinik für Kardiologie und Angiologie, Essen, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: after publication
Access Criteria: contact PI

REFERENCES:
- [Derived] Lortz J, Rassaf T, Jansen C, Knuschke R, Schweda A, Schnaubert L, Rammos C, Koberlein-Neu J, Skoda EM, Teufel M, Bauerle A. A mHealth intervention to reduce perceived stress in patients with ischemic heart disease: study protocol of the randomized, controlled confirmatory intervention "mStress-IHD" trial. Trials. 2023 Sep 15;24(1):592. doi: 10.1186/s13063-023-07618-0. PMID 37715203